CLINICAL TRIAL: NCT04382950
Title: Combination of Recombinant Bacterial ACE2 Receptors -Like Enzyme of B38-CAP and Isotretinoin Could be Promising Treatment for COVID-19 Infection- and Its Inflammatory Complications
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mahmoud Ramadan mohamed Elkazzaz, Sponser Investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COV-2019 Treatment This is
Record Dates: First submitted 2020-05-08; First posted 2020-05-11 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: COVID

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: rbACE2 group plus Aerosolized Isotretinoin (Experimental): rbACE2 0.4 mg/kg IV BID for 7 days (unblinded) plus Aerosolized 13 cis retinoic acid in gradual in 2 divided doses increases froms 0.2 mg/kg/day to 4 mg/kg/day as inhaled 13 cis retinoic acid therapy for 14 days
  Interventions: Combination Product: Recombinant Bacterial ACE2 receptors -like enzyme of B38-CAP (rbACE2) plus Aerosolized 13 cis retinoic acid
- No Intervention: Control group (No Intervention): Standard of care; no placebo

INTERVENTIONS:
Combination Product: Recombinant Bacterial ACE2 receptors -like enzyme of B38-CAP (rbACE2) plus Aerosolized 13 cis retinoic acid — In this study, the experimental group will receive 0.4 mg/kg rbACE2 IV plus Aerosolized 13 cis retinoic acid in gradual in 2 divided doses increases froms 0.2 mg/kg/day to 4 mg/kg/day as inhaled 13 cis retinoic acid therapy for 14 days
  Arms: Experimental: rbACE2 group plus Aerosolized Isotretinoin

SUMMARY:
Combination of Recombinant Bacterial ACE2 receptors -like enzyme of B38-CAP and Isotretinoin could be promising treatment for COVID-19 infection- and Its inflammatory complications

Mahmoud ELkazzaz1

1Department of chemistry and biochemistry, Faculty of Science, Damietta University, Egypt.

_____________________________________________________________________________________________________________________________________________________________________

B38-CAP is a bacteria-derived ACE2-like enzyme that suppresses hypertension and cardiac dysfunction Angiotensin-converting enzyme 2 (ACE2) is critically involved in cardiovascular physiology and pathology, and is currently clinically evaluated to treat acute lung failure. Here we show that the B38-CAP, a carboxypeptidase derived from Paenibacillus sp. B38, is an ACE2-like enzyme to decrease angiotensin II levels in mice. In protein 3D structure analysis, B38-CAP homolog shares structural similarity to mammalian ACE2 with low sequence identity. A study demonstrated that the bacterial B38-CAP as an ACE2-like carboxypeptidase, indicating that evolution has shaped a bacterial carboxypeptidase to a human ACE2-like enzyme. Bacterial engineering could be utilized to design improved protein drugs for hypertension and heart failure. pretreatment of B38-CAP markedly down regulated a massive increase of plasma Ang II levels at 5 min after Ang II injection In addition to the currently used drugs to inhibit Ang II generation or signaling, such as ACE inhibitors or Angiotensin receptor blockers, direct down-modulation of Ang II levels by rhACE2 protein is one of the promising candidates for new therapeutic strategy in cardiovascular disease and other Ang II-related diseases, e.g. ARDS. On the other hand, although mass production of rhACE2 as a protein drug costs due to requirement of mammalian cell expression systems, B38-CAP is easily prepared with E. coli expression system and is cost effective. Therapeutic efficacy and less toxicity in mouse heart failure models would warrant further investigation of B38-CAP or other microbial carboxypeptidases in disease models. Finally the principal investigator expects that treatment with ACE2-like enzyme of bacteria B38-CAP expected to work efficiently Like human ACE2 and it will save the lung cells from COVID - 19 inhibitory effect and down regulation of ACE2 because COVID-19 binds to human ACE2 and down regulates it and this receptors is very important for lung cells survival and function So ,the principal investigator also expects that B38-CAP ACE2 like enzyme may be not recognized by COVID -19 spike protein because evolutionary it is too far away from human ace2 and human ACE2 is a real receptor of COVID -19 not ACE2 like enzyme but in the same time it will make the same function of human ACE2 In another study by Sinha et al who analyzed a publicly available Connectivity Map (CMAP) dataset of pre/post transcriptomic profiles for drug treatment in cell lines for over 20,000 small molecules, isotretinoin was the strongest down-regulator of ACE 2 receptors. On the other hand, they found 6 drugs in CMAP that are currently being investigated in clinical trials for treating COVID-19 (chloroquine, thalidomide, methylprednisolone, losartan, lopinavir and ritonavir, from clinicaltrials.gov), none of which was found to significantly alter ACE2 expression (P>0.1) Moreover, another study demonstrated that isotretinoin is a Potential papain like protease (PLpro) inhibitors which is a protein encoded by SARS-CoV-2 genes and considered one of the proteins that should be targeted in COVID-19 treatment by performing target-based virtual ligand screening . So, the principal investigator expects strong inhibition of COVID - 19 infection And rescuing the lung cells from its serious attack by treating with ACE2 like enzyme and Isotretinoin

Keywords: COVID 2019 , Isotretinoin,B38-CAP , Bacterial ACE2 receptors -like enzyme , rhACE226.

DETAILED DESCRIPTION:
This is a small pilot study investigating whether there is any efficacy signal that warrants a larger Phase 2B trial, or any harm that suggests that such a trial should not be done. It is expected to produce statistically significant results in the major endpoints. The investigator will examine all of the biologic, physiological, and clinical data to determine whether a Phase 2B trial is warranted.

* Primary efficacy analysis will be carried only on patients receiving at least 4 doses of active combination drug. Safety analysis will be carried out on all patients receiving at least one dose of active drug. It is planned to enroll more than or equal to 24 subjects with COVID-19. It is expected to have at least 12 evaluable patients in each group.
* Experimental group: 0.4 mg/kg IV BID for 7 days (unblinded) plus Aerosolized 13 cis retinoic acid in gradual in 2 divided doses increases forms 0.2 mg/kg/day to 4 mg/kg/day as inhaled Isotretinoin therapy for 14 days and standard of care Control group: standard of care Intervention duration: up to 14 days of therapy No planned interim analysis.

Combination of Recombinant Bacterial ACE2 receptors -like enzyme of B38-CAP and Isotretinoin could be promising treatment for COVID-19 infection- and Its inflammatory complications

Mahmoud ELkazzaz1

1Department of chemistry and biochemistry, Faculty of Science, Damietta University, GOEIC, Egypt.

_____________________________________________________________________________________________________________________________________________________________________

Introduction

Angiotensin converting enzyme-2 (ACE2) receptors mediate the entry into the cell of three strains of coronavirus: SARS-CoV, NL63 and SARS-CoV-2. ACE2 receptors are ubiquitous and widely expressed in the heart, vessels, gut, lung (particularly in type 2 pneumocytes and macrophages), kidney, testis and brain. ACE2 is mostly bound to cell membranes and only scarcely present in the circulation in a soluble form. An important salutary function of membrane-bound and soluble ACE2 is the degradation of angiotensin II to angiotensin1-7. Consequently, ACE2 receptors limit several detrimental effects resulting from binding of angiotensin II to AT1 receptors, which include vasoconstriction, enhanced inflammation and thrombosis. The increased generation of angiotensin1-7 also triggers counter-regulatory protective effects through binding to G-protein coupled Mas receptors. Unfortunately, the entry of SARS-CoV2 into the cells through membrane fusion markedly down-regulates ACE2 receptors, with loss of the catalytic effect of these receptors at the external site of the membrane. Increased pulmonary inflammation and coagulation have been reported as unwanted effects of enhanced and unopposed angiotensin II effects via the ACE→Angiotensin II→AT1 receptor axis. Clinical reports of patients infected with SARS-CoV-2 show that several features associated with infection and severity of the disease (i.e., older age, hypertension, diabetes, cardiovascular disease) share a variable degree of ACE2 deficiency. We suggest that ACE2 down-regulation induced by viral invasion may be especially detrimental in people with baseline ACE2 deficiency associated with the above conditions. The additional ACE2 deficiency after viral invasion might amplify the dysregulation between the 'adverse' ACE→Angiotensin II→AT1 receptor axis and the 'protective' ACE2→Angiotensin1-7→Mas receptor axis. In the lungs, such dysregulation would favor the progression of inflammatory and thrombotic processes triggered by local angiotensin II hyperactivity unopposed by angiotensin1-7. In this setting, recombinant brACE2 could be promising therapeutic approaches in patients with SARS-CoV-2 infection.

Rescuing The renin-angiotensin system (RAS) by B38-CAP ACE2 which is a bacteria-derived ACE2-like enzyme

The expected benefits of B38-CAP derived ACE2-like enzyme depending on previous research data show that B38-CAP derived ACE2-like enzyme will do the same function of human ACE2 and in the same time it will be resistant to COVID- spike protein because evolutionary it is too far away from human ace2 and human ACE2 is a real receptor of COVID -19 not ACE2 like enzyme and this discussed as follow :

B38-CAP is a bacteria-derived ACE2-like enzyme that suppresses hypertension and cardiac dysfunction Angiotensin-converting enzyme 2 (ACE2) is critically involved in cardiovascular physiology and pathology, and is currently clinically evaluated to treat acute lung failure. Here we show that the B38-CAP, a carboxypeptidase derived from Paenibacillus sp. B38, is an ACE2-like enzyme to decrease angiotensin II levels in mice. In protein 3D structure analysis, B38-CAP homolog shares structural similarity to mammalian ACE2 with low sequence identity. In vitro, recombinant B38-CAP protein catalyzed the conversion of angiotensin II to angiotensin 1-7, as well as other known ACE2 target peptides. Treatment with B38-CAP suppressed angiotensin II-induced hypertension, cardiac hypertrophy, and fibrosis in mice. Moreover, B38-CAP inhibited pressure overload-induced pathological hypertrophy, myocardial fibrosis, and cardiac dysfunction in mice. Our data identify the bacterial B38-CAP as an ACE2-like carboxypeptidase, indicating that evolution has shaped a bacterial carboxypeptidase to a human ACE2-like enzyme. Bacterial engineering could be utilized to design improved protein drugs for hypertension and heart failure. On the contrary Treatment with recombinant human ACE2 protein (rhACE2), which is devoid of its membrane-anchored domain thus soluble, has been demonstrated to exhibit beneficial effects in various animal models including heart failure, acute lung injury, and diabetic nephropathy, and so forth. rhACE2 is currently tested in the clinic to treat ARDS and COVID-19 infected patients . Using cell cultures and organoids, researchers from the Karolinska Institute in Sweden and the University of British Columbia (UBC) in Canada, showed that by adding a genetically modified variant of ACE2, called human recombinant soluble angiotensin-converting enzyme 2 (hrsACE2), COVID-19 was prevented from entering cells. The paper, published in Cell, shows that hrsACE2 had a dose dependent effect of viral growth of SARS-CoV-2 and was able to reduce it by a factor of 1,000 to 5,000 in cell cultures. Despite its beneficial effects, rhACE2 is a glycosylated protein and thus its preparation requires time- and cost-consuming protein expression system with mammalian or insect cells, which may not be advantageous in drug development and medical economy Although it had been reported that an immune response is associated with the chronic infusion of rhACE2 resulting in the degradation of rhACE226, this was not observed for B38-CAP; there were no antibodies against B38-CAP detectable in the serum of mice infused with B38-CAP for 2 weeks. Implantation of B38-CAP-filled osmotic mini-pumps significantly suppressed Ang II-induced hypertension in conscious mice .without affecting the heart rate. These results indicate that B38-CAP antagonizes the vasopressor effect of Ang II. So the principle investigator expects and suggests that treating with cloned Bacterial ACE2 receptors -like enzyme of B38-CAP could be promising COVID-19 infection- and lung injury preventing drug better than recombinant human ACE2 in addition to brsACE2, expected to lure the virus to attach itself to the copy instead of the actual cells… It distracts the virus from infecting the cells to the same degree and should lead to a reduction in the growth of the virus in the lungs and other organs. A study showed that recombinant B38-CAP protein downregulates Ang II levels in mice and antagonizes Ang II-induced hypertension, pathological cardiac hypertrophy, and myocardial fibrosis. A study showed beneficial effects of B38-CAP on the pathology of pressure overload-induced heart failure in mice without overt toxicities and also pretreatment of B38-CAP markedly downregulated a massive increase of plasma Ang II levels at 5 min after Ang II injection In addition to the currently used drugs to inhibit Ang II generation or signaling, such as ACE inhibitors or Angiotensin receptor blockers, direct down-modulation of Ang II levels by rhACE2 protein is one of the promising candidates for new therapeutic strategy in cardiovascular disease and other Ang II-related diseases, e.g. ARDS. On the other hand, although mass production of rhACE2 as a protein drug costs due to requirement of mammalian cell expression systems, B38-CAP is easily prepared with E. coli expression system and is cost effective. Therapeutic efficacy and less toxicity in mouse heart failure models would warrant further investigation of B38-CAP or other microbial carboxypeptidases in disease models. Furthermore, human ACE2-like enzyme in bacteria might pave the way to a new strategy to engineer evolution of bacterial proteins for better designing and preparations of recombinant protein drugs Finally the principal investigator expect that treatment with ACE2-like enzyme in bacteria B38-CAP may be do the same mechanism of rhACE2 in inhibiting COVID -19 and the other suggested mechanism is that ACE2-like enzyme in bacteria B38-CAP injection in human body will do the same function of human ACE2 and in the same time it will be resistant to COVID- spike protein because evolutionary it is too far away from human ace2 and human ACE2 is a real receptor of COVID -19 not ACE2 like enzyme and Also among three bacterial carboxypeptidases we tested, only B38-CAP showed dependence of proteolytic activity on anion concentration, which is characteristic of ACE2 activity. B38-CAP also showed pH optimum of 7.5 equivalent to rhACE2.In addition, IC50 of MLN-4760 was also equivalent between rhACE2 and B38-CAP. Although B38-CAP exhibited quite similar proteolytic activity to rhACE2, there seems a difference in substrate specificity between two enzymes So , the principal investigator also expects that B38-CAP ACE2 like enzyme may be not recognized by COVID -19 spike protein but in the same time it will make the same function of human ACE2 in addition to down regulating of human ACE2 which is the real receptor of COVID -19

Blocking of ACE2 receptor of COVID -19 which is the real receptors of it

Isotretinoin(13cis RA) may be able to inhibit COVID 2019 entry via down regulation of ACE2 via action like shRNA targeting ACE2 gene expression and this is discussed as follow :

The COVID-19 pandemic caused by SARS-COV-2 has infected over 2,000,000 people causing over 150,000 deaths. A key host cellular protein required for the virus entry is angiotensin-converting enzyme 2 (ACE2) whose expression has been demonstrated in many tissues including alveolar epithelial type II cells in lungs, oral mucosa and intestine, heart, kidney, endothelium and skin. ACE2-expressing cells can act as home cells and are prone to SARS-CoV-2 infection as ACE2 receptor facilitates cellular viral entry and replication. A study demonstrated that patients with hypertension and diabetes mellitus may be at higher risk of SARS-CoV-2 infection, as these patients are often treated with ACE inhibitors (ACEIs) or angiotensin II type-I receptor blockers (ARBs), which have been previously suggested to increase ACE2 expression. In another study by Sinha et al who analyzed a publicly available Connectivity Map (CMAP) dataset of pre/post transcriptomic profiles for drug treatment in cell lines for over 20,000 small molecules, isotretinoin was the strongest down-regulator of ACE 2 receptors. On the other hand, they found 6 drugs in CMAP that are currently being investigated in clinical trials for treating COVID-19 (chloroquine, thalidomide, methylprednisolone, losartan, lopinavir and ritonavir, from clinicaltrials.gov), none of which was found to significantly alter ACE2 expression (P>0.1) Moreover, another study demonstrated that isotretinoin is a Potential papain like protease (PLpro) inhibitors which is a protein encoded by SARS-CoV-2 genes and considered one of the proteins that should be targeted in COVID-19 treatment by performing target-based virtual ligand screening as the Principal Investigator discussed before that (13cRA) is the strongest down-regulator of ACE2. and the principal investigator expects that 13cRA can inhibit and downregulat ACE2 expression ,Suggesting its therapeutic potential in preventing the entry of COVID 2019 to the host cell.

ELIGIBILITY:
Inclusion Criteria:

1.Laboratory diagnosis:

Adult SARI patients with 2019-ncov infection confirmed by PCR; Absolute value of lymphocytes < 0. 6x 109/L; Severe respiratory failure within 48 hours and requires admission to ICU. (severe respiratory failure was defined as PaO2/FiO2 < 200 mmHg and was supported by positive pressure mechanical ventilation (including non-invasive and invasive mechanical ventilation, PEEP>=5cmH2O))

Exclusion Criteria:

* Age <18 years; Age >80 years
* Pregnant or breast feeding woman
* Patient in other therapeutic clinical trial within 30 days before ICF
* Receive any other ACE inhibitors (ACEI), angiotensin-receptor blockers (ARB) treatment within 7 days before ICF
* Chronic immunosuppression: current autoimmune diseases or patients who received immunotherapy within 30 days before ICF
* Hematologic malignancy (lymphoma, leukemia, multiple myeloma)
* Other patient characteristics (not thought to be related to underlying COVID-19) that portend a very poor prognosis (e.g, severe liver failure, and ect)
* Known allergy to study drug or its ingredients related to renin-angiotensin system (RAS), or frequent and/or severe allergic reactions with multiple medications
* Other uncontrolled diseases, as judged by investigators
* Body weight ≥85 kg
* Hypercholesterolemia
* Hypertriglyceridemia
* Liver disease
* Renal disease
* Sjögren syndrome
* Pregnancy
* Lactation
* Depressive disorder
* Contraindications for hormonal contraception or intrauterine device.
* Autoimmune diseases A history of organ, bone marrow or hematopoietic stem cell transplantation
* Patients receiving anti-hcv treatment
* Permanent blindness in one eye
* History of iritis, endophthalmitis, scleral inflammation or retinitis 15-90 days of retinal detachment or eye surgery
* The competent physician considered it inappropriate to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Time course of body temperature (fever) | at 14 days
  Compare the time course of body temperature (fever) between two groups over time.

SECONDARY OUTCOMES:
Viral load over time | 14 days
  Compare viral load between two groups over time.
P/F ratio over time | 14 days
  PaO2/FiO2 ratio
Sequential organ failure assessment score(SOFA score) over time | 14 days
  SOFA, including assessment of respiratory, blood, liver, circulatory, nerve, kidney, from 0 to 4 scores in each systems, the higher scores mean a worse outcome.
Pulmonary Severity Index (PSI) | 14 days
Image examination of chest over time | 14 days
  Based on radiologist's assessment of inflammatory exudative disease, category as follows: significant improvement, partial improvement, no improvement, increase of partial exudation, significant increase in exudation, unable to judge.
Proportion of subjects who progressed to critical illness or death | at 14 days
Time from first dose to conversion to normal or mild pneumonia | 14 days
T-lymphocyte counts over time | 14 days
C-reactive protein levels over time | 14 days
Angiotensin II (Ang II) changes over time | 14 days
Angiotensin 1-7 (Ang 1-7) changes over time | 14 days
Angiotensin 1-5 (Ang 1-5) changes over time | 14 days
Renin changes over time | 14 days
Aldosterone changes over time | 14 days
Angiotensin-converting enzyme (ACE) changes over time | 14 days
Interleukin 6 (IL-6) changes over time | 14 days
Soluble tumor necrosis factor receptor type II (sTNFrII) changes over time | 14 days
Plasminogen activator inhibitor type-1 (PAI-1) changes over time | 14 days
Von willebrand factor (vWF) changes over time | 14 days
Tumor necrosis factor-α (TNF-α) changes over time | 14 days
Soluble receptor for advanced glycation end products (sRAGE) changes over time | 14 days
Surfactant protein-D (SP-D) changes over time | 14 days
Frequency of adverse events and severe adverse events | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: M.Sc. Mahmoud Elkazzaz, M.Sc.Biochemistry, Principal Investigator — General Organization of Export and Import control system